CLINICAL TRIAL: NCT04595734
Title: A Retrospective Study of Clinical Outcomes and Liver-related Toxicity of Patients With Lung Cancer Treated With Immune-checkpoint Inhibitors
Brief Title: Liver Toxicity in Lung Cancer Patients Treated With Immune-checkpoint Inhibitors.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Western Sydney Local Health District (Other)
Collaborators: University of Western Sydney (Other)
Responsible Party: Principal Investigator, Golo Ahlenstiel, Professor of Medicine, Western Sydney Local Health District
Other Study IDs: 2019/PID14816
Record Dates: First submitted 2020-10-14; First posted 2020-10-20 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: Lung Cancer Stage IV; Lung Cancer, Non-small Cell; Hepatitis
Keywords: Immune-checkpoint inhibitors; Lung cancer; Nivolumab; Pembrolizumab; Durvalumab
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Hepatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention due to observational methods of study — No intervention due to observational methods of study

SUMMARY:
Immune-checkpoint inhibitors have recently become available as a new therapy for a variety of cancers. This drugs function by boosting the anti-cancer immune response, but unfortunately, may cause off-target, non-specific immune activation, resulting in liver and gut toxicity. In order to understand the development of liver immune-related adverse events we aim to collect full clinicopathological data from patients with advanced lung cancer treated with immune-checkpoint inhibitors at Blacktown, Westmead and Nepean Hospitals. Patients treated with standard chemotherapy will be used as a control group.

This study aims to establish clinical risk factors that can predict the occurrence of liver immune-related adverse events in patients with advanced lung cancer treated with immune-checkpoint inhibitors. Such predictors may assist in the stratification of patients based on their risk for development liver toxicity as a result of immunotherapy, allowing early cessation/modification of treatment prior to the development of severe adverse reactions. In addition, this retrospective study will aim to determine the significance of pre-existing liver damage on the development of liver adverse events as well as establish a timeline defining the development of adverse events in the liver.

DETAILED DESCRIPTION:
BACKGROUND AND RATIONALE.

Lung cancer is the most common cause of cancer-related mortality worldwide. This year alone 12,817 new lung cancer cases were registered in Australia, the mortality rate of which being 46% within 5 years. Chemotherapy is still considered the first-line treatment, however recent clinical trials have established that with treatment monoclonal antibodies known as immune-checkpoint inhibitors shows higher efficacy in terms of overall survival and progression-free survival. Despite higher efficacy, immune-checkpoint inhibitors can cause a number of immune-related adverse events which may force patients to cease treatment. Among these side effects, liver toxicity occurs rapidly and is asymptomatic in the early stages. These facts underscore the necessity of stratifying patients based on their risk of developing liver toxicity. We aim to predict liver toxicity early on in therapy using data collected from routine clinical testing.

STUDY AIMS / OBJECTIVES.

This retrospective study aims to answer following research questions:

1. Does pre-existing liver fibrosis/cirrhosis influence the development of liver immune-related adverse events?
2. What is the first time-point and subsequent timeline of liver immune-related adverse events occurrence and progression?
3. What clinical markers predict immunotherapy related toxicity?

STUDY DESIGN.

This is non-interventional retrospective study that plans to collect data from patients with stage IV lung cancer treated at Blacktown, Westmead and Nepean Hospitals. The main goal of this study is to establish statistically significant clinical predictors of liver toxicity in patients treated with immune-checkpoint inhibitors. Full clinicopathological data will be collected from hospital medical electronic databases. We will prioritise the examination of liver function blood tests in order to establish the first timepoint of liver function abnormalities and correlate them to pre-treatment blood results.

STUDY PROCEDURES.

This retrospective study will be conducted in 3 steps

1. Collection of full clinicopathological data of patients with advanced lung cancer treated at Blacktown, Westmead and Nepean Hospitals .
2. Blood tests results will be collected according to the following scheme: (1) The day prior to treatment commencement (baseline); (2) every 28th day for patients treated with tyrosine kinase inhibitors; (3) the last day of each therapeutic cycle for patients treated with immune-checkpoint inhibitors or platinum-doublet chemotherapy or combination.
3. Statistical analysis using SPSS v23 and STATA v16 software.

DATA COLLECTION:

1. Clinicopathological data

   * ID
   * Age
   * Sex
   * Clinical diagnosis
   * Histological diagnosis
   * TNM stage
   * Date of diagnosis
   * Date of treatment commencement
   * Therapeutic regimen
   * Cycling regime
   * Date of death
   * Cardiovascular comorbidities
   * Neurologic comorbidities
   * Respiratory comorbidities
   * Endocrine comorbidities
   * Gastrointestinal comorbidities
   * Renal comorbidities
   * Smoking status (pack/years)
   * Eastern Cooperation Oncology Group performance status (ECOG PS)
   * Programmed death ligand 1 (PD-L1) expression (%)
   * Genetic mutations
   * FibroScan data
2. Data from blood tests

   * Red blood cells (RBC)
   * Red blood cells distribution weight (RDW)
   * Haematocrit
   * Haemoglobin
   * Mean corpuscular volume (MCV)
   * Mean corpuscular haemoglobin (MCH)
   * Mean corpuscular haemoglobin concentration (MCHC)
   * Platelets
   * White blood cells (WBC)
   * Neutrophils
   * Lymphocytes
   * Monocytes
   * Eosinophils
   * Basophils
   * Sodium
   * Potassium
   * Bicarbonate
   * Estimated glomerular filtration rate
   * Urea
   * Creatinine
   * Glucose
   * Serum protein
   * Total globulin
   * Albumin
   * Alanine aminotransferase (ALT)
   * Aspartate aminotransferase (AST)
   * Gamma glutamyltransferase (GGT)
   * Alkaline phosphatase (ALP)
   * Total bilirubin
   * C-reactive protein
   * Iron
   * Transferrin
   * Ferritin
3. Statistical considerations:

   * All variables will be analysed using descriptive statistics
   * Mann-Whitney test will be used for estimating differences in liver functional tests between two groups and to evaluate the significance of pre-existing liver damage (counted by APRI and Fib-4 scores) on the development of liver immune-related adverse events
   * Multivariate regression for establishment significant predictors of liver toxicity

ELIGIBILITY:
Inclusion Criteria:

1. - Advanced lung cancer (stage IV)
2. - Treatment - immune-checkpoint inhibitors or chemotherapy
3. - Data is fully available for the whole period of observation

Exclusion Criteria:

1. - Radiologically reported liver metastases
2. - Concurrent treatment with both therapeutic regimes

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with lung cancer treated with immune-checkpoint inhibitors at Blacktown and Westmead Public Hospitals of the Western Sydney Local Health District and Nepean Hospital of the Nepean and Blue Mountains Local Health District.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-01-07 (Actual); Primary Completion 2023-01-10 (Estimated); Study Completion 2025-01-06 (Estimated)

PRIMARY OUTCOMES:
Number of participants with immune-mediated hepatitis | Week 6-12 from treatment commencement
Baseline risk factors significantly correlated with hepatic immune-related adverse events | Week 0
  Blood test results, BMI, FibroScan data will be correlated with the development of liver toxicity

SECONDARY OUTCOMES:
Number of participants with non-hepatic immune-related adverse events | Week 3-32 from treatment commencement
Baseline risk factors significantly correlated with non-hepatic immune-related adverse events | Week 0
  Blood test results and BMI will be correlated with the development of immune-related adverse events (non-hepatic)

CONTACTS AND LOCATIONS:
Overall Officials: Golo Ahlenstiel, Professor, Principal Investigator — Blacktown Hospital, Western Sydney Local Health District
Locations (3):
- Australia (3):
  - Westmead Hospital, Sydney, New South Wales
  - Blacktown Hospital, Sydney, New South Wales
  - Nepean Hospital, Sydney, New South Wales

IPD SHARING:
Plan to Share IPD: Undecided